CLINICAL TRIAL: NCT05224908
Title: Breech Pelvimetry by EOS® Technique With Change of Maternal Position and Delivery Route
Acronym: PelviEOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2021 CHAUVEAU; 2021-A01752-39 (Other: 2021-A01752-39)
Record Dates: First submitted 2021-12-14; First posted 2022-02-04 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: EOS; Pregnancy Related; Fetus Fetus; Breech Fetal Presentation
MeSH Terms: conditions — Fetus-in-Fetu; Breech Presentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pregnant women with a breech fetus (Experimental): pregnant women with a breech fetus performing standing and sitting EOS pelvimetry
  Interventions: Device: EOS

INTERVENTIONS:
Device: EOS — pelvimetry by EOS in standing and sitting position

SUMMARY:
When a patient presents with a fetus in PS after 36+0SA, after acceptance of participation in the study, pelvimetry with evaluation of the height of the fetal presentation by EOS® system in the upright and sitting position will be performed. CT pelvimetry will not be performed. The patient may then be offered an attempt at VME, with clear, fair and appropriate information, after being informed of the data from the right standing EOS® pelvimetry (report and images). VME will be performed according to the recommendations and practice of the department. In the event of failure with a fetus that remains in PS, the choice of delivery route will be decided in consultation with the patient after clear, fair and appropriate information.

If the patient wishes to have a vaginal delivery, the pregnancy will be continued without intervention until spontaneous labour or induction in case of indication (premature rupture of membranes (PMR), over term, or intercurrent maternal or fetal pathology). The modalities of the delivery route and/or a possible induction will be discussed between the obstetric team and the patient.

If the patient wishes a caesarean delivery in case of persistent PS, the delivery will be scheduled after 39+0SA or earlier if indicated (RPM, intercurrent maternal or fetal pathology). In the case of a successful VME with a fetus that remains in cephalic presentation until labour, management will follow current recommendations. The characteristics of the dimensions and angles of the obstetric pelvis and the height of the fetal presentation in the standing and sitting positions, the performance and success of MEC, the choice of delivery route, and the final delivery route will be recorded.

DETAILED DESCRIPTION:
The 3rd trimester ultrasound is performed between 30+0 and 35+0SA, preferably between 30+0 and 32+0SA. In case of breech presentation (PS), an ultrasound check at the Clermont-Ferrand University Hospital from 36+0SA is usually requested. If PS is confirmed, the patient will be given the information sheet concerning breech fetuses published by the Collège National des Gynécologues et Obstétriciens Français (CNGOF) in 2020 and the patient will be offered to participate in the PelviEOS study.

Information about the study will be given by the investigator or his delegates during the presentation ultrasound.

After sufficient time for reflection and consent, EOS® pelvimetry in the upright and sitting position will be performed, starting at 36+0SA, and prior to attempted external manoeuvre version (EMV). The EOS® pelvimetry will be performed in the radiology department of the Clermont-Ferrand University Hospital, Estaing site. No other irradiating examination will be carried out, such as a pelvic CT scan, which will be replaced by pelvimetry using the EOS® system.

The examination will initially be carried out in the standing position, then in the sitting position on a stool.

A marker on the floor represented by two footprints will allow the straight standing and sitting images to be taken with equivalent and reproducible angles of femoral rotation.

The parameters assessed from the images taken by the EOS® system will be in the standing and sitting positions:

* The height of the fetal presentation assessed by measuring the distance between the centre of the maternal bisecting diameter and the lowest fetal trochanter.
* The angle of fetal progression,
* The median transverse diameter (MT),
* Promonto-retro-pubic distance (PRP),
* Magnin's index,
* Measurement of the sacral cord,
* Measurement of the sacral spire,
* Bispinous diameter,
* Bischial diameter,
* Subsacro-subpubic diameter,
* Pelvic angle of incidence,
* Pelvic obliquity,
* coxofemoral angle measurement.

After having been informed of the results of the pelvimetry performed in the upright position only (report and pictures), the performance of a VME will be proposed (the results of the pelvimetry in the sitting position will be transmitted after delivery, for statistical analysis).

If the patient wishes, an attempt at VME in the maternity ward of the Clermont-Ferrand University Hospital can be programmed from 36+0SA in accordance with the recommendations.

In the event of a successful MVA with a fetus that remains in cephalic presentation until labour begins, management will follow current recommendations.

In the event of refusal or failure of VME, the different delivery options will again be explained to the patient in accordance with the recommendations.

If the patient wishes to have a vaginal delivery, the pregnancy will be continued without intervention until spontaneous labour or induction if indicated (premature rupture of membranes (PMR), overdue delivery, intercurrent maternal or fetal pathology). The modalities of the delivery route and/or a possible induction will be discussed between the obstetric team and the patient.

If the patient wishes a caesarean delivery in case of persistent PS, the delivery will be scheduled from 39+0SA or earlier in case of indication (RPM, intercurrent maternal or fetal pathology).

The characteristics of the dimensions and angles of the obstetrical pelvis and the height of the fetal presentation in the standing and sitting positions, the performance and success of a VME, the choice of the delivery route and the actual delivery route will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Major parturient with a breech fetus after 36+0SA.
* Able to give informed consent to participate in the research.
* Enrolled in a Social Security scheme.

Exclusion Criteria:

* Multiple pregnancy
* Pelvimetry by CT scan already performed
* Fetal malformation
* History of pelvic fracture
* Known uterine malformation that precludes VME (unicornuate uterus, uterine septum...)
* Contraindication to vaginal delivery (placenta previa, obstacle previa, bicatric uterus, ...)
* Patient under guardianship or legal protection
* Refusal to participate

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women with a breech fetus
Enrollment: 90 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2025-02-08 (Actual); Study Completion 2025-02-08 (Actual)

PRIMARY OUTCOMES:
Real way of delivery for women with a fetus in PS after 36+0SA. | through the completion of studies, an average of 2 year
  To compare pelvimetry data (different radiographic characteristics of the obstetrical pelvis and height of the fetal presentation (in centimeter) ) recorded by the EOS® system in the standing and sitting positions between cases with a caesarean delivery and cases with a vaginal delivery in pregnant women with a breech fetus after 36+0SA.

SECONDARY OUTCOMES:
Successful completion of the VME | through the completion of studies, an average of 2 year
  To compare pelvimetry data (different radiographic characteristics of the obstetric pelvis and height of fetal presentation (in centimeter)) from the EOS® system in the standing and sitting positions between successful and unsuccessful VME in pregnant women with breech fetuses after 36+0SA.
Intention to deliver vaginally if breech presentation persists | through the completion of studies, an average of 2 year
  To compare pelvimetry data (different radiographic features of the obstetric pelvis and height of fetal presentation (in centimeter)) in pregnant women with breech fetuses after 36+0SA using EOS® in the standing and sitting positions between cases referred for caesarean delivery and cases referred for vaginal delivery.
Measurement of fetal cervical flexion by measuring the craniospinal hinge angle. | through the completion of studies, an average of 2 year
  To study the feasibility of measuring fetal neck flexion (in degrees).

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Chauveau, Study Director — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France